CLINICAL TRIAL: NCT05143203
Title: Evaluation of the Effectiveness of Self-hypnosis on Anxiety and Burnout of Nursing Staff
Acronym: ESHABC
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier Régional Metz-Thionville (Other)
Responsible Party: Sponsor
Other Study IDs: 2021-04Obs-CHRMT
Record Dates: First submitted 2021-11-22; First posted 2021-12-03 (Actual); Last update posted 2023-08-04 (Actual); Status verified 2023-08

CONDITIONS: Hypnosis; Self-hypnosis; Anxiety; Depression; Burn Out
MeSH Terms: conditions — Anxiety Disorders; Depression; Burnout, Psychological

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Staff trained in October 2021: 22 nursing staff will follow two days of Self-Hypnosis training in October 2021
  Interventions: Other: Self-hypnosis training
- Staff trained in May 2021: 22 nursing staff will follow two days of Self-Hypnosis training in May 2021
  Interventions: Other: Self-hypnosis training
- Control staff without training: 22 nursing staff will not follow any training

INTERVENTIONS:
Other: Self-hypnosis training — Self-hypnosis training will be conducted in two phases and the evaluation of effectiveness of the training will be measured using GAD7, PHQ9 and PROQOL questionnaires
  Groups: Staff trained in May 2021; Staff trained in October 2021

SUMMARY:
Its a prospective, non-interventional, single-center study, involving the human person evaluating the impact of self-hypnosis training on anxiety level and burn out in nursing and medical staff

DETAILED DESCRIPTION:
Like other pandemics, that of Covid-19 had a significant psychological impact on the general population. However, this impact turned out to be even more acute among healthcare workers, in connection with repeated exposure to the risk of infection, the reorganization of care and their specific positioning (...) Psychotraumatic, anxiety and depression symptoms has been observed worldwide. The staff of CHR Metz-Thionville were not spared. From the first wave, the caregivers exposed directly to SARS-CoV-2 (emergency, resuscitation, cohorting sector) requested the hypnosis referent doctor of the structure, in order to benefit from hypnosis sessions in order to better manage their anxiety during the sanitary crisis.

The main demand from caregivers was learning stress management tools and a desire for empowerment without psychological support. For information, the support platform set up by the psychiatry service recorded very few calls (39 caregivers from March 24, 2020 to June 26, 2020). Faced with the influx of hypnotherapy requests, the training unit was asked to set up on-site self-hypnosis training.

It seemed important to measure the effect of this learning on the mental health of caregivers using psychometric scales.

This training was initially offered to front-line caregivers in the fight against the covid-19 pandemic and by extension to all caregivers wishing to be trained in this practice.

It is obvious that this pandemic may have worsened a general ill-being of caregivers already present before the current health crisis.

There are many studies on the management of anxiety and pain in patients with a history of chronic disease, and some have focused specifically on learning self-hypnosis techniques. Even if the protocols for learning self-hypnosis techniques are very heterogeneous in these various pathologies, there is a common observation : "studies show positive results on self-esteem, catastrophism, depression, quality of sleep , the somatizations, the anxiety of the patients (and of their parents for the children), mood ".

To date, and to our knowledge, there are no methodologically rigorous studies measuring the effects of hypnosis or self-hypnosis on the mental health of caregivers.

Publications are often limited to clinical cases or positions related to the use of hypnosis and / or self-hypnosis for the well-being of caregivers.

ELIGIBILITY:
Inclusion Criteria:

* Nursing staff of the CHR Metz-Thionville: doctors, nurses or nursing assistants
* Over 18 years old
* Not objecting to participating in the study
* Affiliated to a social security scheme

Exclusion Criteria:

Hospital staff

* Not speaking and/or not understanding the French language.
* Having disorders of higher functions.
* With known history of schizophrenia.
* Deaf or hard of hearing.
* already trained in hypnosis.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Nursing staff: doctors, nurses or nursing assistants
Sampling Method: Non-Probability Sample
Enrollment: 68 (Actual)
Dates: Start 2021-10-12 (Actual); Primary Completion 2022-04-13 (Actual); Study Completion 2023-05-02 (Actual)

PRIMARY OUTCOMES:
Anxiety disorder level evaluation M+6 | 6 months after the training of the training of the first group
  Generalized anxiety disorder screening scale (GAD7) will be measured 6 months after the start of training in self-hypnosis

SECONDARY OUTCOMES:
Anxiety disorder level evaluation D-7 | 7 days before the start of the training of the first group
  Generalized anxiety disorder screening scale (GAD7) The GAD-7 score is calculated by assigning scores of 0, 1, 2, and 3, to the response categories of 'not at all', 'several days', 'more than half the days', and 'nearly every day', respectively, and adding together the scores for the seven questions.
  Scores of 5, 10, and 15 are taken as the cut-off points for mild, moderate and severe anxiety, respectively. When used as a screening tool, further evaluation is recommended when the score is 10 or greater.
Anxiety disorder level evaluation M+1 | 1 month after the start of the training of the first group
  Generalized anxiety disorder screening scale (GAD7) The GAD-7 score is calculated by assigning scores of 0, 1, 2, and 3, to the response categories of 'not at all', 'several days', 'more than half the days', and 'nearly every day', respectively, and adding together the scores for the seven questions.
  Scores of 5, 10, and 15 are taken as the cut-off points for mild, moderate and severe anxiety, respectively. When used as a screening tool, further evaluation is recommended when the score is 10 or greater.
Anxiety disorder level evaluation M+3 | 3 months after the start of the training of the first group
  Generalized anxiety disorder screening scale (GAD7) The GAD-7 score is calculated by assigning scores of 0, 1, 2, and 3, to the response categories of 'not at all', 'several days', 'more than half the days', and 'nearly every day', respectively, and adding together the scores for the seven questions.
  Scores of 5, 10, and 15 are taken as the cut-off points for mild, moderate and severe anxiety, respectively. When used as a screening tool, further evaluation is recommended when the score is 10 or greater.
Anxiety disorder level evaluation M+7 | 7 months after the start of the training of the first group
  Generalized anxiety disorder screening scale (GAD7) The GAD-7 score is calculated by assigning scores of 0, 1, 2, and 3, to the response categories of 'not at all', 'several days', 'more than half the days', and 'nearly every day', respectively, and adding together the scores for the seven questions.
  Scores of 5, 10, and 15 are taken as the cut-off points for mild, moderate and severe anxiety, respectively. When used as a screening tool, further evaluation is recommended when the score is 10 or greater.
Anxiety disorder level evaluation M+12 | 12 months after the start of the training of the first group
  Generalized anxiety disorder screening scale (GAD7) The GAD-7 score is calculated by assigning scores of 0, 1, 2, and 3, to the response categories of 'not at all', 'several days', 'more than half the days', and 'nearly every day', respectively, and adding together the scores for the seven questions.
  Scores of 5, 10, and 15 are taken as the cut-off points for mild, moderate and severe anxiety, respectively. When used as a screening tool, further evaluation is recommended when the score is 10 or greater.
Anxiety disorder level evaluation M+18 | 18 months after the start of the training of the first group
  Generalized anxiety disorder screening scale (GAD7) The GAD-7 score is calculated by assigning scores of 0, 1, 2, and 3, to the response categories of 'not at all', 'several days', 'more than half the days', and 'nearly every day', respectively, and adding together the scores for the seven questions.
  Scores of 5, 10, and 15 are taken as the cut-off points for mild, moderate and severe anxiety, respectively. When used as a screening tool, further evaluation is recommended when the score is 10 or greater.
Depressive disorder evaluation D-7 | 7 days before the start of the training of the first group
  The Patient Health Questionnaire 9-item depression module (PHQ-9) will be used to measure depression disorder of nursing staff 7 days before the start of self-hypnosis training.
  PHQ-9 is a well-validated, brief, self-reported, diagnostic, and severity measure of depression designed for use in primary care.
Depressive disorder evaluation M+1 | 1 month after the start of the training of the first group
  The Patient Health Questionnaire 9-item depression module (PHQ-9) will be used to measure depression disorder of nursing staff 1 month after the start of self-hypnosis training PHQ-9 is a well-validated, brief, self-reported, diagnostic, and severity measure of depression designed for use in primary care.
Depressive disorder evaluation M+3 | 3 months after the start of the training of the first group
  The Patient Health Questionnaire 9-item depression module (PHQ-9) will be used to measure depression disorder of nursing staff 3 months after the start of self-hypnosis training PHQ-9 is a well-validated, brief, self-reported, diagnostic, and severity measure of depression designed for use in primary care.
Depressive disorder evaluation M+6 | 6 months after the start of the training of the first group
  The Patient Health Questionnaire 9-item depression module (PHQ-9) will be used to measure depression disorder of nursing staff 6 months after the start of self-hypnosis training PHQ-9 is a well-validated, brief, self-reported, diagnostic, and severity measure of depression designed for use in primary care.
Depressive disorder evaluation M+7 | 7 months after the start of the training of the first group
  The Patient Health Questionnaire 9-item depression module (PHQ-9) will be used to measure depression disorder of nursing staff 7 months after the start of self-hypnosis training PHQ-9 is a well-validated, brief, self-reported, diagnostic, and severity measure of depression designed for use in primary care.
Depressive disorder evaluation M+12 | 12 months after the start of the training of the first group
  The Patient Health Questionnaire 9-item depression module (PHQ-9) will be used to measure depression disorder of nursing staff 12 months after the start of self-hypnosis training PHQ-9 is a well-validated, brief, self-reported, diagnostic, and severity measure of depression designed for use in primary care.
Depressive disorder evaluation M+18 | 18 months after the start of the training of the first group
  The Patient Health Questionnaire 9-item depression module (PHQ-9) will be used to measure depression disorder of nursing staff 18 months after the start of self-hypnosis training PHQ-9 is a well-validated, brief, self-reported, diagnostic, and severity measure of depression designed for use in primary care.
Professional Quality of Life evaluation D-7 | 7 days before the start of the training of the first group
  The Professional Quality of Life Scale (ProQOL) is a 30 item self-report questionnaire designed to measure compassion fatigue, work satisfaction and burnout in helping professionals. Helping professionals are defined broadly, from those in health care settings, such as psychologists, nurses and doctors. It is useful for workers who perform emotional labour as well as professionals who are exposed to traumatic situations. Raw scores between 10 and 50 are presented for the three subscales (1) Compassion Satisfaction, (2) Burnout and (3) Secondary Traumatic Stress. Each score is also presented as a percentile rank comparing the respondent's scores to scores of helping professionals generally (such as psychologists, doctors, teachers and first responders). A percentile of 50 represents an average score. High scores on Compassion Satisfaction and low scores on Burnout and Secondary Traumatic Stress are indicative of professional health.
Professional Quality of Life evaluation M+6 | 6 Months after the start of the training of the first group
  The Professional Quality of Life Scale (ProQOL) is a 30 item self-report questionnaire designed to measure compassion fatigue, work satisfaction and burnout in helping professionals. Helping professionals are defined broadly, from those in health care settings, such as psychologists, nurses and doctors. It is useful for workers who perform emotional labour as well as professionals who are exposed to traumatic situations. Raw scores between 10 and 50 are presented for the three subscales (1) Compassion Satisfaction, (2) Burnout and (3) Secondary Traumatic Stress. Each score is also presented as a percentile rank comparing the respondent's scores to scores of helping professionals generally (such as psychologists, doctors, teachers and first responders). A percentile of 50 represents an average score. High scores on Compassion Satisfaction and low scores on Burnout and Secondary Traumatic Stress are indicative of professional health.
Professional Quality of Life evaluation M+12 | 12 Months after the start of the training of the first group
  The Professional Quality of Life Scale (ProQOL) is a 30 item self-report questionnaire designed to measure compassion fatigue, work satisfaction and burnout in helping professionals. Helping professionals are defined broadly, from those in health care settings, such as psychologists, nurses and doctors. It is useful for workers who perform emotional labour as well as professionals who are exposed to traumatic situations. Raw scores between 10 and 50 are presented for the three subscales (1) Compassion Satisfaction, (2) Burnout and (3) Secondary Traumatic Stress. Each score is also presented as a percentile rank comparing the respondent's scores to scores of helping professionals generally (such as psychologists, doctors, teachers and first responders). A percentile of 50 represents an average score. High scores on Compassion Satisfaction and low scores on Burnout and Secondary Traumatic Stress are indicative of professional health.
Professional Quality of Life evaluation M+18 | 18 Months after the start of the training of the first group
  The Professional Quality of Life Scale (ProQOL) is a 30 item self-report questionnaire designed to measure compassion fatigue, work satisfaction and burnout in helping professionals. Helping professionals are defined broadly, from those in health care settings, such as psychologists, nurses and doctors. It is useful for workers who perform emotional labour as well as professionals who are exposed to traumatic situations. Raw scores between 10 and 50 are presented for the three subscales (1) Compassion Satisfaction, (2) Burnout and (3) Secondary Traumatic Stress. Each score is also presented as a percentile rank comparing the respondent's scores to scores of helping professionals generally (such as psychologists, doctors, teachers and first responders). A percentile of 50 represents an average score. High scores on Compassion Satisfaction and low scores on Burnout and Secondary Traumatic Stress are indicative of professional health.

CONTACTS AND LOCATIONS:
Overall Officials: Nazmine GULER, MD, Principal Investigator — CHR Metz Thionville Hopital de Mercy
Locations (1):
- Centre Régional Metz-Thionville, Metz, Grand Est, France